CLINICAL TRIAL: NCT06188988
Title: The Interaction Between Viral Infections and the Development of the Airway Microbiome in Young Children With Cystic Fibrosis
Brief Title: Viral Infections and Airway Microbiome in Young Children With Cystic Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: 5812
Record Dates: First submitted 2023-11-09; First posted 2024-01-03 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2023-11

CONDITIONS: Cystic Fibrosis in Children; Respiratory Bacterial Infection; Respiratory Viral Infection; Inflammation Lungs; Respiratory Morbidity
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cystic fibrosis (CF) is the most common hereditary life-threatening condition in Belgium. Because of a dysfunctional cystic fibrosis transmembrane conductance regulator (CFTR) channel, chloride is unable to move to the cell surface and mucus becomes more viscous. Consequently, CF patients are not able to clear their lungs efficiently, and trapped bacteria can lead to chronic infection and inflammation of the lungs, and ultimately respiratory failure.

CF lung disease starts at birth due to muco-inflammatory processes and is associated with a significantly altered microbial colonization of the infant airways compared to infants without CF. Additionally, young children with CF suffer from viral infections as often as their healthy peers, but the episodes are more severe and often prolonged. Moreover, frequent viral infections in children with CF contribute towards a more pathogenic airway microbiome at a young age. Although this link has been previously reported, the exact mechanisms by which this occurs need to be elucidated.

A pulmonary exacerbation in CF is characterized by an increase in respiratory symptoms, general symptoms and a decline in lung function. Most young children with CF suffer from a mean of 4 exacerbations per year for which antibiotics are prescribed. Despite the current novel therapies in CF, treatment of respiratory infections stay relevant and is a greater challenge with increasing survival.

The key objective of this study is to gain insights into the mechanisms by which viral infections leading to pulmonary exacerbations induce a more pathogenic microbiome in young children with CF.

About forty participants will be recruited at the paediatric CF clinic of the Antwerp University Hospital. Inclusion criteria are an age of less than 5 years and a diagnosis of CF. There are no exclusion criteria. Duration of the study is 1 year to cover for seasonality of clinical symptoms. Study visits are scheduled at 3-month intervals corresponding with the regular follow up, or unscheduled during an acute pulmonary exacerbation. From all participants, two oropharyngeal swabs (for microbiome analysis and for immunological/mucin analysis) will be collected at set time points. For the linking of the laboratory data to the clinical characteristics, we will examine demographics, environmental exposures, and disease markers of CF. Next to the collection of the oropharyngeal swabs, a history, physical examination, and technical investigations will be performed at the study visits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis

Exclusion Criteria:

* None

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be recruited at the paediatric cystic fibrosis clinic of the Antwerp University Hospital. Inclusion criteria are an age of less than 5 years and a diagnosis of cystic fibrosis (confirmed by sweat chloride levels > 60 mmol/L and/or two pathogenic CFTR variants).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
airway microbial profiles of young cystic fibrosis patients | 1 year
  Metagenomic shotgun sequencing after extraction of bacterial DNA from oropharyngeal swabs
airway inflammatory profiles of young cystic fibrosis patients | 1 year
  cytokine levels in oropharyngeal swabs, measured by multiplex ELISA
Airway mucin profiles of young cystic fibrosis patients | 1 year
  mucin profiles in oropharyngeal samples via qRT-PCR
Demographic data of young cystic fibrosis patients | 1 year
  Age (in years), CFTR genotype (description of mutation), Sex (male/female), ethnicity (hispanic or latino/not hispanic or latino), race (american indian or alaska native/asian/black or african american/native hawaiian or other pacific islander/white)
Environmental data in young cystic fibrosis patients | 1 year
  Mode of birth delivery (vaginal delivery / caesarian section), birth weight (in kg), feeds in infancy (breastfeeding exclusively/breastfeeding in combination with formula/exclusively formula feeding), smoke exposure (prenatal/postnatal/ongoing), day care (Yes/No), vaccinations (according to schedule/not according to schedule), physical activity (Yes/No), parent education (mother normal or low level, father normal or low level), household income (normal/low level), postcode (number), rural living (yes/no), urban living (Yes/no), season of sampling (spring/summer/autumn/winter), type of medication (name), duration of medication (in weeks), type of antibiotics for pulmonary exacerbation (name), duration time of antibiotics for pumonary exacerbation (in weeks)
Disease markers of young cystic fibrosis patients | 1 year
  RR (in /min), SpO2 ( in %), BMI (in kg/m2), temperature (in °C), rhinosinusitis (yes/no), nasal congestion (yes/no), acute otitis media (yes/no), fever (yes/no), decreased activity level (yes/no), dyspnea (Yes/no), cough (Yes/no), sputum production (yes/no), wheezing (yes/no), crackles (yes/no), differential air entry (yes/no), bronchiolitis (yes/no), pneumonia (yes/no), pulmonary exacerbation (yes/no), CFQ-R score, lung function FEV1 (Z-score), lung function LCI (Z-score), bronchiectasis on CT scan (yes/no), wall thichening on CT scan (Yes/no), mucous plugging on CT scan (yes/no), air trapping on CT scan (Yes/No), previously or new relevant (extra)pulmonary conditions/illnesses (name of diagnoses)

SECONDARY OUTCOMES:
Virome profiling in young cystic fibrosis patients during an acute pulmonary exacerbation | 1 month
  Extensive profiling of viruses in young cystic fibrosis patients after taking orpharyngeal sample during an acute pulmonary exacerbation by multiplex qPCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No